CLINICAL TRIAL: NCT03633383
Title: Outcomes of Transcatheter Aortic Valve Implantation in Management of Severe Symptomatic Aortic Stenosis
Acronym: TAVI
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Moustafa Mohamed, Assistant Lecturer, Assiut University
Other Study IDs: 17200225; 1906 (Other: Assiut Univeristy Faculty of Medicine Ethical Committee)
Record Dates: First submitted 2018-07-14; First posted 2018-08-16 (Actual); Last update posted 2018-08-16 (Actual); Status verified 2018-08

CONDITIONS: Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Transfemoral Approach
  Interventions: Device: Transcatheter aortic valve
- Transapical Approach
  Interventions: Device: Transcatheter aortic valve

INTERVENTIONS:
Device: Transcatheter aortic valve — Self-expandable aortic valve prothesis

SUMMARY:
TAVI is still a relatively new technique that is emerging with advance in the percutaneous and implantable valve technology. Despite its safe use in inoperable and high risk patients with severe symptomatic aortic valve stenosis, minimizing complications, predictors of outcomes and approach preference is still an area of study. Here we decided to study the outcomes of patients undergoing TAVI, different approaches used and their subsequent results and complications.

DETAILED DESCRIPTION:
Severe symptomatic aortic stenosis in elderly patients represents a surgical challenge for cardiac surgeons due to heavy calcifications and associated comorbidities. Such conditions usually are associated with dramatic intra and postoperative complications leading to many cases being declined for open surgical replacement. Many treatment modalities were described including trans-catheter valvotomy but with only temporary improvements and high rates of recurrence.

Transcatheter Aortic Valve Implantation (TAVI) has offered an alternative solution to such cases in which open surgery is deemed too risky or prohibited. Percutaneous Heart Valves (PHV) implantations have been experimented on animals since the early 1990s. Yet the first human case was not reported till 2002, in which a percutaneously implanted heart valve (PHV) composed of 3 bovine pericardial leaflets mounted within a balloon-expandable stent was developed and implanted through the antegrade trans-septal approach in a patient presenting with severe calcific aortic stenosis associated with many noncardiac comorbidities including leg ischaemia. Despite Patient's death after 17 weeks due to noncardiac causes, his follow-up showed significant improvement of left ventricle (LV) function and aortic valve area after implantation of the percutaneous valve.

This case was followed by several single-center and small multicenter registries and series that included inoperable or very-high-risk patients, which were associated with promising results that confirmed the feasibility of TAVI.

Many approaches are used for TAVI with the transfemoral approach being the primary option. Abnormalities of the iliofemoral anatomy have led to the emergence of other approaches including transapical, subclavian, axillary, and transaortic routes. Potential advantages of such approaches would be the avoidance of using large catheters though the iliofemoral system, aortic arch, ascending aorta, and aortic valve. Yet, their main disadvantage would be the need for general anaesthesia.

As any surgical procedure, TAVI carries some risk of complications, major vascular injuries, stroke, conduction abnormalities, myocardial infarction, coronary obstruction and acute kidney injury have been reported. Although, careful planning, patient selection, perioperative workup and individualised approach choice play an important role in avoiding such problems.

ELIGIBILITY:
Inclusion Criteria:

* Patients with severe symptomatic aortic stenosis undergoing TAVI.

Exclusion Criteria:

* Patients with concomitant valvular heart disease.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who meet the listed inclusion and exclusion criteria will be eligible for the study
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-08-31 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
All cause mortality | one month
  Causes of mortality such stroke, myocardial infarction, kidney injury,bleeding

SECONDARY OUTCOMES:
Stroke | One month
  Major or minor
Myocardial infarction | One month after tavi
Bleeding | One month after tavi
  Amount of blood loss post Tavi
Hospital stay | One month
  Calculated in days
Acute kidney injury | One month
  According to RIFLE system
Number of patients with conduction disturbance and pacemaker implantation | 6 months
  AV block by Electrocardiogram
Gradient on implanted valve | One month
  By echocardiography measured in mmhg
Degree of transvalvular leakage | One month
  By echocardiography divided in no, mild, moderate and severe

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Ghoneim, Professor, Study Chair — Assiut University; Hussien Elkhayat, Lecturer, Study Director — Assiut University

REFERENCES:
- [Background] Andersen HR, Knudsen LL, Hasenkam JM. Transluminal implantation of artificial heart valves. Description of a new expandable aortic valve and initial results with implantation by catheter technique in closed chest pigs. Eur Heart J. 1992 May;13(5):704-8. doi: 10.1093/oxfordjournals.eurheartj.a060238. PMID 1618213
- [Background] Cribier A, Eltchaninoff H, Bash A, Borenstein N, Tron C, Bauer F, Derumeaux G, Anselme F, Laborde F, Leon MB. Percutaneous transcatheter implantation of an aortic valve prosthesis for calcific aortic stenosis: first human case description. Circulation. 2002 Dec 10;106(24):3006-8. doi: 10.1161/01.cir.0000047200.36165.b8. PMID 12473543
- [Background] Rodes-Cabau J. Transcatheter aortic valve implantation: current and future approaches. Nat Rev Cardiol. 2011 Nov 15;9(1):15-29. doi: 10.1038/nrcardio.2011.164. PMID 22083020
- [Background] Chow SC, Cheung GS, Lee AP, Wu EB, Ho JY, Kwok MW, Yu PS, Wan IY, Underwood MJ, Wong RH. Transcatheter aortic valve implantation: the transaortic approach. Asian Cardiovasc Thorac Ann. 2017 Jun;25(5):357-363. doi: 10.1177/0218492317702027. Epub 2017 May 17. PMID 28513189
- [Background] Tamburino C, Capodanno D, Ramondo A, Petronio AS, Ettori F, Santoro G, Klugmann S, Bedogni F, Maisano F, Marzocchi A, Poli A, Antoniucci D, Napodano M, De Carlo M, Fiorina C, Ussia GP. Incidence and predictors of early and late mortality after transcatheter aortic valve implantation in 663 patients with severe aortic stenosis. Circulation. 2011 Jan 25;123(3):299-308. doi: 10.1161/CIRCULATIONAHA.110.946533. Epub 2011 Jan 10. PMID 21220731
- [Background] Masson JB, Kovac J, Schuler G, Ye J, Cheung A, Kapadia S, Tuzcu ME, Kodali S, Leon MB, Webb JG. Transcatheter aortic valve implantation: review of the nature, management, and avoidance of procedural complications. JACC Cardiovasc Interv. 2009 Sep;2(9):811-20. doi: 10.1016/j.jcin.2009.07.005. PMID 19778768